CLINICAL TRIAL: NCT04898738
Title: Prospective COVID-19 Cohort Study to Assess the Epidemiology, Transmission and Control of SARS-CoV-2 in the Dominican Republic
Brief Title: Prospective COVID-19 Cohort Study, Dominican Republic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); London School of Hygiene and Tropical Medicine (Other); The University of Queensland (Other); Yale University (Other); Broad Institute of MIT and Harvard (Other); Ministerio de Salud Publica y Asistencia Social, Republica Dominicana (Other Government)
Responsible Party: Principal Investigator, Eric J. Nilles, M.D.,M.S.C., Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2021p001294
Record Dates: First submitted 2021-05-19; First posted 2021-05-24 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: SARS-CoV-2 Infection; Covid19
MeSH Terms: conditions — COVID-19 | interventions — Ethanol

STUDY DESIGN:
Intervention Model Description: This is a prospective cohort study that aims to prospectively monitor 2,000 community-based study participants with serial serological screening for SARS-CoV-2 and enhanced molecular surveillance for active infection. Nested within this cohort is a randomized trial that will allocate study participants into two arms: thoe that receive versus do not receive alcohol-based hand sanitizer (ABHS) through the course of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alcohol-based hand sanitizer (Active Comparator): Half the study households with receive ABHS through the course of the study
  Interventions: Other: Alcohol based hand sanitizer
- No Alcohol-based hand sanitizer (No Intervention): Half the study households with not receive ABHS through the course of the study

INTERVENTIONS:
Other: Alcohol based hand sanitizer — Provision of ABHS to randomly selected households
  Arms: Alcohol-based hand sanitizer

SUMMARY:
This project will build on an existing CDC funded cooperative agreement in the Dominican Republic with the Brigham and Women's Hospital (2018-2023) that includes (i) prospective COVID-19 and AFI surveillance at two health facilities and (ii) a nationally representative cross-sectional community-based serological survey of approximately 7,000 healthy adults and children targeting SARS-CoV-2 and other AFI pathogens to be conducted between April and June 2021. This linked study will establish a nested cohort of 2,000 participants enrolled in the national serological survey and prospectively monitor them for COVID-19 symptoms, conduct serial serological testing, implement molecular surveillance for SARS-CoV-2 and sequencing for variants of concern, implement and evaluate WASH mitigation measures, and monitor uptake and perceptions of COVID-19 vaccines.

ELIGIBILITY:
Inclusion Criteria:

* Previously enrolled in a linked national community-based seroepidemiological study in the Dominican Republic
* Agreed and consented to be recontacted to participate in additional research studies at the time of enrollment in #1
* ≥2 years of age
* Agree to participate

Exclusion Criteria:

* Ward of the State

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1043 (Actual)
Dates: Start 2021-08-18 (Actual); Primary Completion 2022-11-22 (Actual); Study Completion 2023-02-10 (Actual)

PRIMARY OUTCOMES:
Hand hygiene practices | 1 year
  The average daily frequency of study participant hand hygiene events over the previous seven days will be assessed using standardized survey questionnaires at 0-, 3-, 6-, 9-, and 12-months.

SECONDARY OUTCOMES:
Acceptability of hand hygiene technology | 1 year
  Study participants preference for different hand hygiene technology (e.g. soap and water, ABHR) as measured using a five-point Likert Scale at 0-, 3-, 6-, 9-, and 12-months.
SARS-Cov-2 seroconversion | 1 year
  Number of study participants that seroconvert from SARS-CoV-2 seronegative to seropositive at time points 0-, 6-, and 12-months as assessed by presence of anti-nucleocapsid immunoglobulin

CONTACTS AND LOCATIONS:
Overall Officials: Eric J Nilles, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Community study, Santo Domingo, Dominican Republic

IPD SHARING:
Plan to Share IPD: Yes
De-identified data for epidemiological analyses and modelling (including demographic data, clinical data, and survey questionnaire survey) will be shared with the following collaborators: Adam Kucharski (LSHTM), Colleen Lau (University of Queensland), Marietta Vasquez (Yale University), Matt Lozier (US CDC), Pardis Sabeti (Broad Institute), and staff at the Health Ministry Division of Epidemiology. Non-identifiable data shared with listed collaborators will be performed with secure file transfer.